CLINICAL TRIAL: NCT05054504
Title: Integration of Butterfly iQ Point of Care Ultrasound Into Antenatal Care in Blantyre, Malawi: A Feasibility and Acceptability Study
Brief Title: Feasibility and Acceptability of Butterfly iQ
Acronym: FAB-IQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jhpiego (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Johns Hopkins Bloomberg School of Public Health (Other); Kamuzu University of Health Sciences (Other); Ministry of Health, Malawi (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ARC-005
Record Dates: First submitted 2021-09-04; First posted 2021-09-23 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Pregnancy Related
Keywords: Butterfly IQ; Malawi; Blantyre; Antenatal care; ANC/PNC Research Collective; Point of care ultrasound; Bill & Melinda Gates Foundation; Johns Hopkins Research Project; Johns Hopkins Bloomberg School of Public Health

STUDY DESIGN:
Intervention Model Description: The primary intervention under study is the Butterfly iQ ultrasound, embedded in a larger program of training, iterative service delivery design, and a final program evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intervention (Other): The primary intervention is a multi-phase, mixed methods, implementation research study that will investigate the feasibility and acceptability of the limited introduction of ultrasound via the Butterfly iQ device into routine ANC service delivery at health center level in Blantyre, Malawi. The study will occur in three phases: 1) Training, 2) Iterative Service Delivery, and 3) Final Evaluation.
  Interventions: Device: Butterfly iQ

INTERVENTIONS:
Device: Butterfly iQ — The primary intervention under study is the Butterfly iQ point-of-care ultrasound device, embedded in a larger program of training, iterative ANC service delivery design, and a final program evaluation.

SUMMARY:
The purpose of this study is to investigate feasibility and acceptability of a novel intervention to integrate Butterfly IQ into antenatal care (ANC) service delivery in Malawi. The study will also explore potential impact of the intervention on selected service delivery outcomes and identification of abnormal pregnancies.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the feasibility and acceptability of a novel intervention to integrate Butterfly IQ into ANC service delivery in Blantyre, Malawi. This study will further the understanding of antenatal ultrasound in Malawi by testing the following hypothesis:

When planned and implemented collaboratively with local stakeholders, limited introduction and integration of point-of-care ultrasound with Butterfly iQ into ANC service delivery at health center level will be feasible and acceptable for health providers and clients.

The study intervention will include a multi-phased approach to design, introduction, improvement, and evaluation of Butterfly IQ for routine obstetric ultrasound integrated into ANC service delivery in Malawi.

Phase 1: Training Phase 1 includes training on Butterfly IQ, integration in ANC workflow, and referral/counter-referral within network.

Phase 2: Iterative Service Delivery Phase 2 includes weekly evaluation and iterative re-design of services.

Phase 3: Final Evaluation Phase 3 includes evaluation for potential integration into current policies and frameworks; determination to pursue pending additional factors; or determination of incompatibility, as well as selected support for transition/handover, if applicable.

ELIGIBILITY:
Eligibility criteria by phase and participant type

Phase 1 Inclusion Criteria

1. Member of HC or hospital staff providing obstetric care.
2. Able and willing to comply with all study requirements and complete all study procedures.
3. Able and willing to provide informed consent to be screened for and to take part in the study.

Phase 1 Exclusion Criteria 1. Has any condition that, in the opinion of the investigator/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Phase 2 Inclusion Criteria

Study Participant - Health Center and Hospital Staff:

1. Member of HC or hospital staff providing obstetric care.
2. Able and willing to comply with all study requirements and complete all study procedures.
3. Able and willing to provide informed consent to be screened for and to take part in the study.

Study Participant - ANC Clients:

Participants must meet all criteria to be eligible for inclusion in the study:

1. Age 18 years or older at Screening, as verified per site Standard Operating Procedures (SOPs).
2. At enrollment, present for first ANC visit.
3. Able and willing to comply with all study requirements and complete all Phase 2 study procedures.
4. Able and willing to provide informed consent to be screened for and to take part in Phase 2 of the study.
5. Intention to stay within study catchment area for study Phase 2 duration and willingness to give adequate locator information, as defined in site SOPs.

Phase 2 Exclusion Criteria

Study Participant - Health Center and Hospital Staff:

1. Has any condition that, in the opinion of the investigator/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Study participant - ANC Clients:

1. Has any condition that, in the opinion of the investigator/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Phase 3 Inclusion Criteria

1. Participated in Phase 1 or 2 of the study or newly recruited stakeholder interested in development or implementation of obstetric ultrasound in Malawi.
2. Able and willing to comply with all study requirements and complete all Phase 3 study procedures.
3. Able and willing to provide informed consent to be screened for and to take part in Phase 3 of the study.

Phase 3 Exclusion Criteria

1. Has any condition that, in the opinion of the investigator/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1575 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Feasibility of the intervention by participant report | 7 months
  Proportion of enrolled midwives who report the intervention to be feasible
Feasibility of the intervention by quality standards met (ultrasound) | 7 months
  Proportion of ultrasound examinations found to meet quality standards
Feasibility of the intervention by quality standards met (ANC) | 7 months
  Proportion of ANC visits (that included Butterfly IQ) found to meet quality standards
Feasibility of the intervention by observation of functioning systems | 7 months
  Proportion of Butterfly IQ systems functioning at end of study period
Feasibility of the intervention by observation of environments of care | 7 months
  Proportion of participating HC with facilitative environments of care

SECONDARY OUTCOMES:
Acceptability, by participant report (providers) | 7 months
  Proportion of providers who find the intervention acceptable
Acceptability, by participant report (ANC clients) | 7 months
  Proportion of ANC clients who find the intervention acceptable

OTHER OUTCOMES:
Gestational age at first ANC contact | 7 months
  Median gestational age at first ANC contact
Number and types of suspected and confirmed higher-risk conditions identified by ultrasound and recorded in study records | 7 months
  Numbers of the following
  * Ectopic pregnancy
  * Multiple gestation
  * Abnormal placentation
  * Intrauterine fetal demise
  * Abnormalities of amniotic fluid, e.g., oligohydramnios, polyhydramnios
  * Fetal anomaly
  * Other condition not specified above

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Noguchi, PhD, MSN, Study Director — Jhpiego, Johns Hopkins University; Linly Seyama, Principal Investigator — University of Malawi College of Medicine, JHP Blantyre
Locations (1):
- Johns Hopkins Research Project, Blantyre, Malawi